CLINICAL TRIAL: NCT03279848
Title: Stratification of Stroke Rehabilitation: 5-year Profiles of Functional Outcomes
Status: Completed | Type: Observational
Sponsor: Tai Po Hospital (Other Government)
Responsible Party: Principal Investigator, Bryan Ping Ho CHUNG, Principal Investigator of Physiotherapy Department, Tai Po Hospital
Other Study IDs: 2016.283
Record Dates: First submitted 2017-08-31; First posted 2017-09-12 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Stroke Rehabilitation
MeSH Terms: interventions — Stroke Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:  — Stroke rehabilitation
  Other Names: Stroke Rehabilitation

SUMMARY:
Objective: To make use of admission Modified Functional Ambulation Category (MFAC) as a stratification tool to reveal profiles of functional outcomes of patients with stroke in inpatient rehabilitation.

Design: This was a retrospective, descriptive study of the demographic, functional outcomes of patients with stroke in an inpatient rehabilitation centre. A total of 2,722 patients completed a stroke rehabilitation program from 2011 to 2015 were recruited.

DETAILED DESCRIPTION:
Objective: To make use of admission Modified Functional Ambulation Category (MFAC) as a stratification tool to reveal profiles of functional outcomes of patients with stroke in inpatient rehabilitation.

Design: This was a retrospective, descriptive study of the demographic, functional outcomes of patients with stroke in an inpatient rehabilitation centre. A total of 2,722 patients completed a stroke rehabilitation program from 2011 to 2015 were recruited. The patients were divided into seven groups according to their admission Modified Functional Ambulation Category (MFAC). The between-group difference in length of stay (LOS), functional outcomes at admission and discharge including Modified Rivermead Mobility Index (MRMI) and Modified Barthel Index (MBI) as well as MRMI gain, MRMI efficiency, MBI gain and MBI efficiency were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with principal diagnosis of cerebrovascular accident, stroke, or hemiplegia and has received and completed stroke rehabilitation program in a hospital in Hong Kong between the periods of 1st January 2011 to 31st December 2015.

Exclusion Criteria:

* Patients with principal diagnosis of cerebrovascular accident, stroke, or hemiplegia and has received but cannot completed stroke rehabilitation program in a hospital in Hong Kong between the periods of 1st January 2011 to 31st December 2015.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with principal diagnosis of cerebrovascular accident, stroke, or hemiplegia.
Sampling Method: Non-Probability Sample
Enrollment: 2722 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Modified Rivermead Mobility Index (MRMI) | baseline and 1 month
  MRMI was used to assess subjects' mobility in this study. The MRMI is highly reliable between raters (ICC= 0.98) and has high internal consistency (Cronbach's alpha = 0.93) to early stage patients with stroke. The MRMI consists of eight test items, including turning over, changing from lying to sitting, maintaining sitting balance, going from sitting to standing, standing, transferring, walking indoors, and climbing stairs. The score of MRMI range from 0 to 40. One main characteristic of the MRMI is that participants are scored by observation of their performance on the items directly. Change in MRMI i.e. MRMI gain is the difference between pre-discharge MRMI and admission MRMI.

SECONDARY OUTCOMES:
Change in Modified Barthel Index (MBI) Gain | baseline and 1 month
  MBI was used to assess subjects' basic activities of daily living (ADL) in this study. MBI measures the subject's performance on ten functional items including self-care, continence, and locomotion. The values assigned to each item are based on the amount of physical assistance required to perform the task and added to give a total score ranging from 0 to 100 (0 = fully dependent, 100 = fully independent) with higher score indicating higher levels of physical function. There are no subtotal score because there are no sub-scales. The internal consistency reliability coefficient for MBI is 0.90. Change in MBI i.e. MBI gain is the difference between pre- discharge MBI and admission MBI.